CLINICAL TRIAL: NCT04988048
Title: Collaborative Study to Evaluate Heterologous Vaccination Against Covid-19 in Argentina
Acronym: ECEHeVac
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Public Health, Argentina (Other Government)
Collaborators: Russian Direct Investment Fund (Industry)
Responsible Party: Principal Investigator, Marina Pasinovich, md, Medical adviser on immunizations, Undersecretary of Health Strategies, Ministry of Public Health, Argentina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0001/2021
Record Dates: First submitted 2021-07-29; First posted 2021-08-03 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: COVID-19 VACCINE; Covid19
Keywords: Interchangeability; Heterologous vaccination
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; Gam-COVID-Vac vaccine; BIBP COVID-19 vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Randomized, open, multicenter, collaborative and adaptive non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Gam-COVID-Vac C1/ ChAdOx1 nCoV-19 (Active Comparator): Heterologous: Gam-COVID-Vac C1/ ChAdOx1 nCoV-19
  Interventions: Biological: COVID-19 vaccines
- ChAdOx1 nCoV-19 / Gam-COVID-Vac C1 (Active Comparator): Heterologous: ChAdOx1 nCoV-19 / Gam-COVID-Vac C1
  Interventions: Biological: COVID-19 vaccines
- Gam-COVID-Vac C1/ BBIBP-CorV (Active Comparator): Heterologous: Gam-COVID-Vac C1/ BBIBP-CorV
  Interventions: Biological: COVID-19 vaccines
- BBIBP-CorV / Gam-COVID-Vac C1 (Active Comparator): Heterologous: BBIBP-CorV / Gam-COVID-Vac C1
  Interventions: Biological: COVID-19 vaccines
- ChAdOx1 nCoV-19 / BBIBP-CorV (Active Comparator): Heterologous: ChAdOx1 nCoV-19 / BBIBP-CorV
  Interventions: Biological: COVID-19 vaccines
- BBIBP-CorV / ChAdOx1 nCoV-19 (Active Comparator): Heterologous: BBIBP-CorV / ChAdOx1 nCoV-19
  Interventions: Biological: COVID-19 vaccines
- Gam-COVID-Vac C1/ mRNA-1273 (Active Comparator): Heterologous: Gam-COVID-Vac C1/ mRNA-1273
  Interventions: Biological: COVID-19 vaccines
- ChAdOx1 nCoV-19 / mRNA-1273 (Active Comparator): Heterologous: ChAdOx1 nCoV-19 / mRNA-1273
  Interventions: Biological: COVID-19 vaccines
- BBIBP-CorV / mRNA-1273 (Active Comparator): Heterologous BBIBP-CorV / mRNA-1273
  Interventions: Biological: COVID-19 vaccines
- Gam-COVID-Vac C1/ Gam-COVID-Vac C2 (Active Comparator): Homologous: Gam-COVID-Vac C1/ Gam-COVID-Vac C2
  Interventions: Biological: COVID-19 vaccines
- ChAdOx1 nCoV-19 / ChAdOx1 nCoV-19 (Active Comparator): Homologous: ChAdOx1 nCoV-19 / ChAdOx1 nCoV-19
  Interventions: Biological: COVID-19 vaccines
- BBIBP-CorV / BBIBP-CorV (Active Comparator): Homologous: BBIBP-CorV / BBIBP-CorV
  Interventions: Biological: COVID-19 vaccines
- mRNA-1273 / mRNA-1273 (Active Comparator): Homologous: mRNA-1273 / mRNA-1273
  Interventions: Biological: COVID-19 vaccines
- Gam-COVID-Vac C1/ Gam-COVID-Vac C1 (Active Comparator): Homologous: Gam-COVID-Vac C1/ Gam-COVID-Vac C1
  Interventions: Biological: COVID-19 vaccines

INTERVENTIONS:
Biological: COVID-19 vaccines — Gam-COVID-Vac Gamaleya National Center for Epidemiology and Microbiology - Russia. Non-replicative viral vector. Multi-dose vial (5 doses in 3 mL) Single-dose vial (1 dose in 0.5 mL). Intramuscular T° less than -18 ° C
  BBIBP-CorV Beijing Institute of Biological Products - People's Republic of China. Inactivated viruses. Single-dose vials (1 dose in 0.5 mL) or multi-dose vial (2 doses per vial). Intramuscular T° 2 to 8 ° C
  ChAdOx1 nCoV-19 vaccine AZD1222 AstraZeneca-Oxford - United Kingdom. Non-replicative viral vector. Multi-dose vial (10 doses in 5 mL). Intramuscular T°: 2 to 8 ° C
  mRNA-1273 or Spikevax Moderna Switzerland GmbH and the National Institute of Allergy and Infectious Diseases (NIAID) of the United States. mRNA. Multi-dose vial (maximum 15 doses per 0.5ml vial). Intramuscular. T°-15 ° to -50 °
  Other Names: SPUTNIK-V (Gam-COVID-Vac); SINOPHARM (BBIBP-CorV); AstraZeneca (ChAdOx1 nCoV-19 vaccine AZD1222); Moderna (mRNA-1273 or Spikevax)

SUMMARY:
Randomized, open, multicenter, collaborative and adaptive non-inferiority trial to evaluate the immunogenicity and reactogenicity of the heterologous vaccination schedules made up of the combination of vaccines available in Argentina (Sputnik-V, AstraZeneca, Sinopharm and Moderna); and to compare the immunogenicity and reactogenicity of heterologous and homologous vaccination schedules.

DETAILED DESCRIPTION:
More than a hundred COVID-19 vaccines based on different technologies are currentlyin the clinical phase of development around the world. More than a dozen derived from different platforms have been approved by regulatory entities in several countries and are used to immunize the world's population.

The dynamics of the COVID-19 pandemic, the emergence of variants, the magnitude and durability of the immune response, the effectiveness of approved vaccination schemes, as well as the possibility of combining vaccines from various platforms, are some of the issues to be facedin public health decision-making, in order to deliver the best protection standards to the population.

Given the dynamics of the disease in Argentina, the access to different COVID-19 vaccination alternatives requires the development of various strategies, such as stratifying the population sampled by the risk of being infected or transmitting the disease, the agreement for the acquisition of vaccines produced by multiple laboratories simultaneously, setting as a priority first dose vaccination to a higher number of people in a shorter period of time and completing the schemes already started.

The pandemic has revealed the capacity of our country to carry out research studies that produce evidence to face the new challenges posed by COVID19 and, particularly,to implement vaccination as one of the main tools to reduce the health impact it generates-for example,six months after the start of the vaccination campaign, results demonstrate the positive impact of this strategy and its effectiveness.

Models based on heterologous immunization schemes with vaccines from different platforms require evaluation by means of clinical trials,in order to show whether they are not less effective than homologous schemes already established. This is achieved through comparative evaluation of their immunogenicity, efficacy and reactogenicity with studies considering implementation possibilities, adaptiveness and response to real life situations.

Hence, the Ministry of Health propoundsthe development of a collaborative network for the integration of studies on vaccination strategies against COVID-19 with the use of heterologous schemes based on the evaluation of their non-inferiority, compared to homologous vaccination schedulesalready implemented worldwide.

The Argentine Ministry of Health looks forward to generating solid scientific evidence that supports decision-making in health policies, with broad federal participation and common objectives.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, vaccinated with 1 dose of Sputnik V, AstraZeneca or Sinopharm vaccine up to 60 days prior to enrollment (according to the platform of the vaccine received as the first dose) or not vaccinated for the mRNA-1273 / mRNA-1273 Arm
* With and without identified risk factors for COVID-19
* Signature of the informed consent
* Remain in the jurisdiction where your study began until the end of it
* Be able to understand and sign the informed consent

Exclusion Criteria:

* Patients with immunocompromise due to underlying disease or immunosuppressive treatment
* Pregnant and breastfeeding people
* Being registered in the National Health Surveillance System for having suffered COVID-19 (symptomatic or asymptomatic) or having a positive IgG result in nucleocapsid ELISA in the sample taken on "DAY 0" for people who had received Sputnik-V or AstraZeneca as the first dose
* Having had a severe allergic reaction (anaphylaxis) to any vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1760 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Antibody against Spike protein measurement by ELISA test | 28 days
  To assess IgG anti Spike response (UI/ml): To assess the antibody concentration in each arm by ELISA COVIDAR IgG expressed in IU/ml. To determine whether a heterologous vaccination regimen is non-inferior to that observed with currently used homologous regimens.
Incidence of adverse events by measurement of the number of reactions after vaccination | 28 days
  Adverse events events presumably attributable to vaccination and immunization (ESAVI) and adverse events of special interest (AESI)

SECONDARY OUTCOMES:
Neutralising Antibody against Spike protein and cellular immune response | 6 month
  Neutralizing antibody titer in the serum of vaccinated individuals, using "Vero" cells as infection targets and cellular immune response It will be studied in heparinized blood samples using mononuclear cells isolated from the blood samples obtained. These cells will be challenged "in vitro" with "pools" of peptides from the Spike and N proteins of SARS-CoV-2, evaluating the production of the cytokines interferon-γ and IL-2 by T cells, by flow cytometry.
Incidence of adverse events by measurement of the number of reactions after vaccination | 6 months
  adverse events events presumably attributable to vaccination and immunization (ESAVI) and adverse events of special interest (AESI)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Pasinovich, MD, Principal Investigator — Ministry of Public Health, Argentina
Locations (4):
- Argentina (4):
  - Córdoba, Córdoba
  - Provincia de Buenos Aires, La Plata
  - La Rioja, La Rioja
  - San Luis, San Luis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nunez NG, Schmid J, Power L, Alberti C, Krishnarajah S, Kreutmair S, Unger S, Blanco S, Konigheim B, Marin C, Onofrio L, Kienzler JC, Costa-Pereira S, Ingelfinger F; InmunoCovidCba; InViV working group; Pasinovich ME, Castelli JM, Vizzotti C, Schaefer M, Villar-Vesga J, Mundt S, Merten CH, Sethi A, Wertheimer T, Lutz M, Vanoaica D, Sotomayor C, Gruppi A, Munz C, Cardozo D, Barbas G, Lopez L, Carreno P, Castro G, Raboy E, Gallego S, Moron G, Cervi L, Acosta Rodriguez EV, Maletto BA, Maccioni M, Becher B. High-dimensional analysis of 16 SARS-CoV-2 vaccine combinations reveals lymphocyte signatures correlating with immunogenicity. Nat Immunol. 2023 Jun;24(6):941-954. doi: 10.1038/s41590-023-01499-w. Epub 2023 Apr 24. PMID 37095378